CLINICAL TRIAL: NCT06486298
Title: Comparison Between Vacuum Drain and Passive Drain In Abdominoplasty : Randomized Clinical Study
Brief Title: Comparison Between Vacuum Drain and Passive Drain In Abdominoplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Pola Fayez Fanos, plastic surgery departement, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Soh-Med-23-12-10MS
Record Dates: First submitted 2024-03-19; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Abdominoplasty Surgery
Keywords: abdominoplasty surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vacuum Drain insertion at abdominoplasty surgery (Active Comparator): insert the active drain after adominoplasty with radivac container
  Interventions: Device: Vacuum Drain and Passive Drain insertion at abdominoplasty surgery
- Passive Drain insertion at abdominoplasty surgery (Experimental): insert the passive drain after adominoplasty with collecting bag
  Interventions: Device: Vacuum Drain and Passive Drain insertion at abdominoplasty surgery

INTERVENTIONS:
Device: Vacuum Drain and Passive Drain insertion at abdominoplasty surgery — Compare the subcutaneous collection with Vacuum Drain and Passive Drain insertion at abdominoplasty surgery

SUMMARY:
The aim of the present study is to:

Compare the subcutaneous collection with Vacuum Drain and Passive Drain insertion at abdominoplasty surgery

ELIGIBILITY:
Inclusion Criteria:

* • Cooperative male and female patients aged between 20-60 years old.

  * All patients in the study presented with varying degrees of excess abdominal skin and adipose tissue, along with a range of underlying abdominal muscle laxity, following volumetric changes of the abdominal cavity.
  * These patients may undergo after bariatric surgery, dietry weight loss or after multiple pregnancies.

Exclusion Criteria:

* • Uncooperative patients unwilling to give consent.

  * Those unsuitable for abdominoplasty surgery, BMI >30 and those on antiplatelet medication.
  * Unfit for surgery and patients with allergies to any of the anesthesia components.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
the subcutaneous collection with vaccum drain | 10 days
  the subcutaneous collection with Vacuum Drain at abdominoplasty surgery regarding : Incidence of postoperative complications
the subcutaneous collection with passive drain | 10 days
  the subcutaneous collection with passive Drain at abdominoplasty surgery regarding : Incidence of postoperative complications

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag Hospital University, Sohag, Egypt